CLINICAL TRIAL: NCT01669369
Title: A Prospected Randomized Multicenter Clinical Trial of Lithium Carbonate Combined With Neo-adjuvant Chemotherapy to Treat Osteosarcoma
Brief Title: Clinical Trial of Lithium Carbonate Combined With Neo-adjuvant Chemotherapy to Treat Osteosarcoma
Acronym: Li2CO3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Nanfang Hospital, Southern Medical University (Other); Shenzhen Second People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lithium-5010
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Osteosarcoma
Keywords: Lithium Carbonate; Chemotherapy; prognosis
MeSH Terms: conditions — Osteosarcoma | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The shape,color and smell of placebo are similar to Lithium Carbonate tablet used in the treatment arm.Patients in this arm take placebo twice a day.
  Interventions: Drug: Placebo
- Lithium Carbonate (Experimental): Patients in this arm take Lithium Carbonate twice a day with a dose of 20-25mg/kg/d.
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — 400 patients were randomly divided into two groups according to sequence of entering the group: lithium carbonate group and control group (1:1). Patients in lithium carbonate group were treated with combinations of chemotherapy and lithium carbonate, the control group were treated with chemotherapy only. Patients were suggesting continuing this trial until the end of the chemotherapy regimen or being confirmed as disease progression by RECIST.
  Other Names: Lithobid
  Arms: Lithium Carbonate
Drug: Placebo — The shape,color and smell of placebo are similar to Lithium Carbonate tablet used in the treatment arm.Patients in this arm take placebo twice a day.
  Other Names: PLACEBO TREATMENT
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Lithium Carbonate combined with neo-adjuvant chemotherapy improve the prognosis of osteosarcoma

DETAILED DESCRIPTION:
Osteosarcoma is the most common primary malignant bone tumor in childhood and adolescence, the prognosis for the disease is poor. What's more, chemotherapy resistance and serious myelosuppression occur frequently in clinical further hindered canonical adjuvant chemotherapy. In our previous researches, we observed that GSK-3B positively regulates the NF-kB pathway to promote proliferation and tumorigenicity in osteosarcoma cell. Targeted inhibition of GSK3beta showed an obvious antitumor effect. It is a promising therapeutic target in osteosarcoma, especially if GSK-3b inhibition is combined with chemotherapeutic drugs. Lithium carbonate, commonly use in clinical application because of its fine quality and cheap price, was proven to be effected as a kind of GSK3beta inhibitor and stimulating factor of peripheral blood leukocyte. Therefore, lithium carbonate theoretically possesses effects of both anti-tumor as well as improvement of myelosuppression. We look forward to the results of clinical trials to test the effect of combinations of chemical drugs with lithium carbonate on myelosuppression, disease-free survival rate and lung metastasis rate in patients with osteosarcoma who treated with conventional chemotherapeutic regimens and wide resection. This study is a multi-centre, double-blind, randomized clinical trial phase 4. The inclusion criterion is patients with primary osteosarcoma in femur, tibia and humerus（IIB）. With the help of statistic method, 400 patients were randomly divided into two groups according to sequence of entering the group: lithium carbonate group and control group (1:1). Patients were suggesting continuing this trial until the end of the chemotherapy regimen or being confirmed as disease progression by RECIST guiding principles. According to their histological types, patients are analyzed using subgroup analysis. Disease evaluation will be conducted every 8 weeks. A follow-up to count the overall survival rate after grouping was performed within at least 24 months or at most 120 months. Our study may represent a novel and feasible approach by combination of conventional chemotherapy drugs and targeted drugs. More importantly, it may hopefully be a promising strategy to improve overall survival of osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed primary classical osteosarcoma in extremities
* staging IIB
* MRI showing no skip lesion
* receive standard neo-adjuvant chemotherapy, adjuvant chemotherapy,and standard surgical treatment

Exclusion Criteria:

* a history of non-standard treatment(chemotherapy or surgery)
* secondary osteosarcoma or well-differentiated parosteal osteosarcoma
* evident dysfunction of cardia,liver and kidney, or pregnant women or women during lactation

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival,incidence of chemotherapy-induced myelosuppression | at least 24 months or at most 120 months

SECONDARY OUTCOMES:
over-all survival,metastasis-free survival | at least 24 months or at most 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The first affiliated hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Because our research has not yet finished, we would decide whether or not make individual participant data (IPD) available to other researchers according to the result of this study.

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903